CLINICAL TRIAL: NCT03497676
Title: Phase I/II Study of the Safety, Acceptability, Tolerability, and Pharmacokinetics of Oral and Long-Acting Injectable Cabotegravir and Long-Acting Injectable Rilpivirine in Virologically Suppressed HIV-Infected Children and Adolescents
Brief Title: More Options for Children and Adolescents (MOCHA): Oral and Long-Acting Injectable Cabotegravir and Rilpivirine in HIV-Infected Children and Adolescents
Acronym: MOCHA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2017; 30070 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1C: CAB (Experimental): Step 1: CAB administered orally as one 30 mg tablet once daily, beginning at the Entry visit, for 4-6 weeks.
  Step 2 (Q4W dosing): CAB LA administered as three single intramuscular (IM) injections four weeks apart (600 mg injection at Week 4b, 400 mg injection at Week 8, and 400 mg injection at Week 12).
  Step 2 (Q8W dosing): CAB LA administered as two single IM injections four weeks apart (600 mg injection at Week 4b and 600 mg injection at Week 8).
  Interventions: Drug: Oral Cabotegravir (CAB); Drug: Long-Acting Injectable Cabotegravir (CAB LA); Drug: Combination Antiretroviral Therapy (cART)
- Cohort 1R: RPV (Experimental): Step 1: RPV administered orally as one 25 mg tablet once daily, beginning at the Entry visit, for 4-6 weeks.
  Step 2 (Q4W dosing): RPV LA administered as three single IM injections four weeks apart (900 mg injection at Week 4b, 600 mg injection at Week 8, 600 mg injection at and Week 12).
  Step 2 (Q8W dosing): RPV LA administered as two single IM injections four weeks apart (900 mg injection at Week 4b and 900 mg injection at Week 8).
  Interventions: Drug: Oral Rilpivirine (RPV); Drug: Long-Acting Injectable Rilpivirine (RPV LA); Drug: Combination Antiretroviral Therapy (cART)
- Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA (Experimental): Step 3: CAB administered orally as one 30 mg tablet once daily and RPV administered orally as one 25 mg tablet once daily, beginning at the Entry visit for 4-6 weeks.
  Step 4: First and second injections: CAB LA administered as a 600 mg IM injection and RPV LA administered as a 900 mg IM injection at Week 4b and at Week 8. Subsequent injections: starting at Week 16, CAB LA administered as a 600 mg IM injection and RPV LA administered as a 900 mg IM injection every eight weeks through Week 96 or final safety extension visit.
  Interventions: Drug: Oral Cabotegravir (CAB); Drug: Oral Rilpivirine (RPV); Drug: Long-Acting Injectable Cabotegravir (CAB LA); Drug: Long-Acting Injectable Rilpivirine (RPV LA)
- Cohort 2B: CAB LA + RPV LA (Experimental): Step 5: First and second injections: CAB LA administered as a 600 mg IM injection and RPV LA administered as a 900 mg IM injection at Entry and at Week 4. Subsequent injections: starting at Week 12, CAB LA administered as a 600 mg IM injection and RPV LA administered as 900 mg IM injection every eight weeks through Week 92 or final safety extension visit.
  Interventions: Drug: Long-Acting Injectable Cabotegravir (CAB LA); Drug: Long-Acting Injectable Rilpivirine (RPV LA)

INTERVENTIONS:
Drug: Oral Cabotegravir (CAB) — 30 mg tablets administered orally
  Arms: Cohort 1C: CAB; Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Drug: Oral Rilpivirine (RPV) — 25 mg tablets administered orally
  Other Names: Edurant
  Arms: Cohort 1R: RPV; Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Drug: Long-Acting Injectable Cabotegravir (CAB LA) — Administered by intramuscular (IM) injection
  Arms: Cohort 1C: CAB; Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA; Cohort 2B: CAB LA + RPV LA
Drug: Long-Acting Injectable Rilpivirine (RPV LA) — Administered by intramuscular (IM) injection
  Arms: Cohort 1R: RPV; Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA; Cohort 2B: CAB LA + RPV LA
Drug: Combination Antiretroviral Therapy (cART) — Participants continued their pre-study cART regimen. The antiretroviral drugs in participants' cART regimens were not provided through the study.
  Arms: Cohort 1C: CAB; Cohort 1R: RPV

SUMMARY:
The purpose of this study was to determine the dosage for oral cabotegravir (CAB) and long-acting cabotegravir (CAB LA) and long-acting rilpiverine (RPV LA) and evaluate the safety, acceptability, tolerability, and pharmacokinetics (PK) of oral CAB, CAB LA, and RPV LA in virologically suppressed children and adolescents living with HIV.

DETAILED DESCRIPTION:
IMPAACT 2017 was a Phase I/II, multi-center, open-label, non-comparative dose-finding study with the primary objective of evaluating the safety, acceptability, tolerability, and PK of oral cabotegravir (CAB) and long-acting cabotegravir (CAB LA) as well as long-acting rilpivirine (RPV LA) in adolescents living with HIV-1, who are 12 to <18 years of age, ≥35kg, and virologically suppressed.

The study design included two cohorts of participants and five study steps. In Cohort 1, Step 1 participants received either oral CAB or oral rilpivirine (RPV) for at least four weeks and up to six weeks (maximum). In Cohort 1, Step 2 participants received intramuscular injectable formulations of the study products, either CAB LA or RPV LA. Cohort 1 participants were assigned either CAB (Cohort 1C) or RPV (Cohort 1R) based on their pre-study combination Antiretroviral Therapy (cART) regimen. Participants on a PI-based and/or NNRTI-based cART regimen were assigned to Cohort 1C, and participants on a non-boosted INSTI-based cART regimen were assigned to Cohort 1R. All participants continued their pre-study cART regimen during Cohort 1.

During Cohort 2, all participants discontinued their pre-study cART regimen and received both study products, CAB and RPV, at the doses established in Cohort 1. Cohort 2 participants enrolled to either Cohort 2A to receive both oral CAB + oral RPV (Step 3) followed by both CAB LA + RPV LA (Step 4) or Cohort 2B to directly receive both CAB LA + RPV LA without an oral lead-in phase (Step 5). If eligible, Cohort 1 participants were able to enroll into Cohort 2 (i.e., Cohort 1 Rollover). However, Cohort 2 participants who were not previously enrolled in Cohort 1 (i.e., Cohort 1-Naïve) were the primary group for analyses and conclusions. No participants enrolled into Cohort 2B, direct to injection (Step 5). Therefore, all references to Cohort 2 refer to Cohort 2A (Steps 3 and 4).

Two interim analyses were planned. The first interim analysis established the doses for Cohort 2 and determined whether to open Cohort 2 to Cohort 1 participants who met criteria to enter Cohort 2. The second interim analysis provided justification to open Cohort 2 to additional participants who were not previously enrolled in Cohort 1. A final analysis of Cohort 1 data was performed to confirm the final doses for Cohort 2.

Safety and PK evaluations were performed during Steps 1-5 and long-term safety follow-up (LSFU). Antiviral activity assessments were performed during Steps 1-5. Acceptability and tolerability were assessed during Steps 1-5 and LSFU, with all participants completing quantitative questionnaires and a subset of participants completing in-depth qualitative interviews. Additionally, parents/caregivers of a subset of U.S. participants from U.S. sites were also enrolled to complete a single in-depth qualitative interview. Because objectives related to parents/caregivers were exploratory, these outcomes are not described here.

Cohort 1 participants were followed for up to 64 weeks. Participants were followed for at least four weeks in Step 1 (oral phase) and at least 12 weeks in Step 2 (injection phase). All Step 2 participants were followed (on cART, off study product) for up to an additional 48 weeks as part of LSFU after their last study product injection. If eligible, Cohort 1 participants enrolled into Cohort 2 before completing LSFU. For Cohort 1, Step 1 participants not progressing to Step 2, the last visit was targeted to be completed 28 days after the participant's last oral study product use.

Cohort 2 participants were followed for up to 188 (Cohort 2B) or 192 (Cohort 2A) weeks. Participants were followed for at least four weeks in Step 3 (oral phase) and 92 weeks in Step 4/Step 5 (injection phase). After completing 92 weeks of follow-up in Step 4/Step 5 (injection phase), Cohort 2 participants who continued access to injectable study products through a mechanism external to the protocol exited the study. If it was not possible for participants to access injections of CAB LA + RPV LA from non-study sources at the completion of their Step 4 Week 96 or Step 5 Week 92 visit, participants remained in the study safety extension for up to 48 weeks. Participants who permanently discontinued injectable study product use during Cohort 2, Step 4/Step 5, or did not wish to continue to access the study products through the external mechanism after their Week 96 visit, were followed (on cART, off study product) for an additional 48 weeks as part of LSFU after their last study product injection, except for participants in the study safety extension. Participants in the study safety extension who decided to permanently discontinue injectable study product or who had not established access to study product after the 48 weeks in the study safety extension would exit the study (not enter LSFU). For Cohort 2, Step 3 participants not progressing to the injection phase, the last visit was targeted to be completed 28 days after the participant's last oral study product use. Female participants who discontinued study product use (either oral or injectable study product) due to pregnancy during Steps 1-5 were followed for an additional 48 weeks in LSFU to assess long-term safety and washout PK of the study products, except for participants in the study safety extension. Participants who became pregnant during the safety extension were only followed until the pregnancy outcome was determined.

ELIGIBILITY:
Inclusion Criteria: Cohort 1 Step 1, Cohort 2 Step 3, and Cohort 2 Step 5

All the following criteria must be met for inclusion of any adolescent participant in Step 1 of Cohort 1, or in Step 3 of Cohort 2, unless otherwise noted:

* At enrollment, body weight greater than or equal to 35 kg (77 lbs)

  * Note: For Cohort 1 Step 2 participants, body weight will not be exclusionary for enrollment into Cohort 2 Step 3, if otherwise eligible.
* For Cohort 1, at enrollment, body mass index (BMI) less than or equal to 31.5 kg/m^2
* At enrollment, willing and able to comply with the study visit schedule and other study requirements, as determined by the site investigator or designee
* Confirmed HIV-1-infection based on documented testing of two samples collected at different time points. More information on this criterion can be found in the protocol.
* For at least 3 consecutive months (defined as 90 consecutive days) prior to screening, and prior to enrollment, has been on stable unchanged cART consisting of 2 or more drugs from 2 or more classes of antiretroviral drugs, ascertainment of this criterion may be based on parent or guardian report only, but available medical records should also be reviewed in relation to this criterion.

  * Note: Participants undergoing dose modifications to their antiretroviral regimen for growth or who are switching medication formulation(s) are considered to be on a stable cART.
* Has at least one documented plasma HIV-1 RNA less than the lower limit of detection of the assay from a specimen collected 6 to 12 months (defined as 180 to 365 days) prior to entry. OR

Has at least one documented plasma HIV-1 RNA less than the lower limit of detection of the assay from a specimen collected less than 6 months (defined as within 179 days) prior to entry and at least one documented plasma HIV-1 RNA result less than the lower limit of detection of the assay from a specimen collected in the 12-18 months (defined as 365 to 545 days) prior to entry.

OR

For Cohort 1 participants enrolling to Cohort 2, has documented plasma HIV-1 RNA results less than the lower limit of detection of the assay from all indicated Cohort 1 study visits with their Cohort 1 Week 16 visit completed within 28 days prior to Cohort 2 entry.

* At screening, has Grade 2 or lower of all the following laboratory test results:

  * Alanine transaminase (ALT) (u/l)
  * Lipase (u/l)
  * Estimated creatinine clearance (CrCl; Schwartz formula mL/min/1.73m^2)
  * Platelets (cells/mm^3)
  * Hemoglobin (g/dL)
  * AST (u/l)
  * Absolute Neutrophil Count (cells/mm3)
  * See study protocol for guidance on severity grading. Laboratory tests may be repeated during the study screening period, with the latest result used for eligibility determination.
* At screening, is on an atazanavir-containing (ATV) cART regimen, and has total bilirubin less than or equal to 1.5 mg/dL or normal direct bilirubin
* At screening, has documented plasma HIV-1 RNA less than 50 copies/mL
* At screening, mean value of Q-T interval (QTc) interval (automated machine readout or calculated using either Bazett or Fredericia) on ECG performed in triplicate, less than or equal to 500 msec.
* For females, has a negative (blood or urine) human chorionic gonadotropin (hCG) laboratory test result at entry
* For females of childbearing potential, at entry, currently using at least one allowable effective method of contraception, and agrees to use at least one allowable effective method of contraception throughout study participation, for at least 30 days after discontinuation of oral study product, and for at least 48 weeks after discontinuation of CAB LA and/or RPV LA, and intending to delay any planned pregnancies until 30 days after last oral study product use or until 48 weeks after last injectable study product use.

  * Note: See study protocol for details regarding contraceptive counseling, a list of the allowed effective contraceptive methods for this study, and the definition of a female of childbearing potential. Hormonal-based contraceptives must have been initiated within the prescribed time, per the respective contraceptive method, to be considered effective at the time of Entry. The site IoR or designee is responsible for ensuring that the contraceptive is used in accordance with the approved product label, and counseling participants on proper use of chosen methods of contraception, including barrier methods.
* For Cohort 1 participants enrolling to Cohort 2, have completed all scheduled product injections and completed Week 16 visit in Cohort 1 Step 2

Exclusion Criteria: Cohort 1 Step 1, Cohort 2 Step 3, or Cohort 2 Step 5

Adolescents will be excluded from the study if any of the following are identified during the screening period:

* Within 6 months (defined as within 179 days) prior to entry, two consecutive documented HIV-1 RNA values greater than the lower limit of detection of the assay

  * Note: Unconfirmed virologic HIV-1 RNA value of greater than the lower limit of detection of the assay (transient detectable viremia, or "blip") prior to screening is not exclusionary.
* For Cohort 1 participants enrolling to Cohort 2, Step 3, occurrence of any Grade 3 or higher adverse event assessed as related to study product or permanent discontinuation of study product due to an adverse event of any grade assessed as related to study product during participation in Cohort 1 (including any long-term safety and washout PK follow-up visits).
* For participants enrolling to Cohort 1 Step 1, based on available medical records, currently on either a cART regimen containing both a protease inhibitor (PI) and an integrase strand transfer inhibitor (INSTI), or a cART regimen containing both an INSTI and a non-nucleoside reverse transcriptase inhibitor (NNRTI).
* As determined by the IoR or designee, and based on available medical records, known or suspected resistance to RPV
* As determined by the IoR or designee based on available medical records, known or suspected resistance to INSTIs
* History of congestive heart failure, symptomatic arrhythmia, or any clinically significant cardiac disease, as determined by the IoR or designee based on available medical records
* At entry, known active tuberculosis infection, requiring anti-tuberculosis treatment, as determined by the IoR or designee based on available medical records
* Known hepatitis B or hepatitis C infection, as determined by the IoR or designee based on available medical records
* Clinically significant hepatic disease, as determined by the IoR or designee based on available medical records
* Current or anticipated need for chronic anti-coagulation, as determined by the IoR or designee, based on available medical records
* History of sensitivity to heparin or heparin-induced thrombocytopenia, as determined by the IoR or designee, based on available medical records
* History of known or suspected bleeding disorder including history of prolonged bleeding, as determined by the IoR or designee, based on available medical records
* Known or suspected allergy to study product components
* More than one seizure within one year (defined as within 365 days) prior to entry, or unstable or poorly controlled seizure disorder, as determined by the IoR or designee, based on available medical records.
* At entry, participant is receiving (or has received in the last 7 days) any disallowed medication listed in the study protocol.
* Current inflammatory skin condition that compromises the safety of intramuscular injections as determined by the IoR or designee.
* Has a tattoo or other dermatological condition overlying the buttock region which, in the opinion of the IoR or designee, may interfere with interpretation of injection site reactions
* Surgically-placed, or planned, buttock implants, per self-report
* For females, lactating (per self-report and/or parent/guardian report) at entry
* Enrolled in another clinical trial of an investigational agent, device, or vaccine
* Any other condition or social circumstance situation that, in the opinion of the IoR or designee, would make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Inclusion/Exclusion Criteria, Step 2 (Cohort 1 Progression Criteria, Step 1 to Step 2)

Cohort 1 Step 1 participants will be assessed for eligibility to progress from the oral lead-in phase (Step 1) to the injection phase (Step 2) primarily based on the safety assessments from the Cohort 1 Step 1 Week 4a study visit. Clinical assessments conducted prior to administering the first injection at the Week 4b visit will also be used to confirm eligibility to receive the injectable study product. See the study protocol for Week 4a and Week 4b visit scheduling, order of procedures, and visit windows, respectively.

All of the following criteria must be met in order for participants to be included in Cohort 1 Step 2:

* Currently enrolled in Cohort 1, Step 1
* At Cohort 1 Step 1 Week 4a study visit, or from confirmatory repeat testing of Cohort 1 Step 1 Week 4a study visit laboratory tests, has Grade 2 or lower of all the following laboratory test results:

  * ALT (u/l)
  * Lipase (u/l)
  * Estimated creatinine clearance (CrCl; Schwartz formula mL/min/1.73m^2)
  * Platelets (cells/mm^3)
  * Hemoglobin (g/dL)
  * AST (u/l)
  * Absolute Neutrophil Count (cells/mm3)
  * Note: For a Grade 2 ALT test result from this visit, refer to the study protocol for required participant management. Abnormal laboratory test result values from the Week 4a visit may be repeated within the target visit window, and if confirmatory testing results in Grade 2 or lower, the participant may be eligible to continue onto the injection phase, should all other eligibility criteria be met.
* For females, at Cohort 1 Step 1 Week 4b study visit, has a negative hCG laboratory test result
* Assessed by the IoR or designee as sufficiently adherent in Step 1 to permit an adequate evaluation of safety and tolerability as part of the oral lead-in phase prior to entry into the injection phase
* Participants who meet any of the following criteria will be excluded from Cohort 1 Step 2:

  * Has permanently discontinued oral study product
  * Occurrence of any grade 3 or higher adverse event assessed as related to study product during participation in Step 1
  * Any other condition or social circumstance that, in the opinion of the IoR or designee, would make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Inclusion/Exclusion Criteria, Step 4 (Cohort 2 Progression Criteria, Step 3 to Step 4)

Cohort 2 Step 3 participants will be assessed for eligibility to progress from the oral lead-in phase (Step 3) to the injection phase (Step 4) primarily based on the safety assessments from the Cohort 2 Step 3 Week 4a study visit. Clinical assessments conducted prior to administering the first injection at the Week 4b visit will also be used to confirm eligibility to receive the injectable study product. See the study protocol for Week 4a and Week 4b visit scheduling, order of procedures, and target visit windows, respectively.

All of the following criteria must be met in order for participants to be included in Cohort 2 Step 4:

* Currently enrolled in Cohort 2, Step 3
* At Cohort 2 Step 3 Week 4a study visit, or from confirmatory repeat testing of Cohort 2 Step 3 Week 4a study visit laboratory tests, has Grade 2 or lower of the following laboratory test results:

  * ALT (u/l)
  * Lipase (u/l)
  * Estimated creatinine clearance (CrCl; Schwartz formula mL/min/1.73m^2)
  * Platelets (cells/mm^3)
  * Hemoglobin (g/dL)
  * AST (u/l)
  * Absolute Neutrophil Count (cells/mm3)
  * Note: For a Grade 2 ALT test result from this visit, refer to the study protocol for required participant management. Abnormal laboratory test result values from the Week 4a visit may be repeated, within the target visit window, and if confirmatory testing results in Grade 2 or lower, the participant may be eligible to continue onto the injection phase, should all other eligibility criteria be met.
* For females, at Cohort 2 Step 3 Week 4b study visit, has a negative hCG laboratory test result
* Assessed by the IoR or designee as sufficiently adherent in Step 3 to permit an adequate evaluation of safety and tolerability as part of the oral lead-in phase prior to entry into the injection phase
* Participants who meet any of the following criteria will be excluded from Cohort 2 Step 4:

  * Has permanently discontinued oral study products
  * Occurrence of any grade 3 or higher adverse event assessed as related to study product during participation in Cohort 2, Step 3
  * Any other condition or social circumstance that, in the opinion of the IoR or designee, would make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Inclusion/Exclusion Criteria: Parents/Caregivers

Selected parents or caregivers of adolescents may be enrolled to complete qualitative phone interviews. See the study protocol for more information regarding the selection process, and coordination of scheduling the interviews. All of the following criteria must be met for the parent/caregiver to be enrolled:

* Selected by the protocol team for participation in the study
* Willing and able to provide informed (verbal or written) consent for study participation
* Per the adolescent participant, has knowledge of how the adolescent participant tolerated the study product, and lives with or has regular supportive contact with the adolescent participant
* Per parent/caregiver self-report, has knowledge of how the participant tolerated the study product, and lives with or has regular supportive contact with the adolescent participant
* Willing and able to complete interview in English by phone
* Parents and/or caregivers of participants who meet the following criterion will be excluded from study participation:

  * Any condition or social circumstance that, in the opinion of the IoR or designee, would make study participation unsafe for either the parent/caregiver or the adolescent participant, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bolton Moore, MSc, MBBCh, Study Chair — Centre for Infectious Disease Research in Zambia/University of Alabama Birmingham; Aditya H. Gaur, MD, Study Chair — St. Jude Children's Research Hospital
Locations (19):
- United States (8):
  - Usc La Nichd Crs, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Pediatric Perinatal HIV NICHD CRS, Site 5127, Miami, Florida
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Baylor College of Medicine/ Texas Children's Hospital NICHD CRS, Houston, Texas
- Botswana (2):
  - Gaborone CRS, Gaborone, South-East District
  - Molepolole CRS, Site 12702, Molepolole
- South Africa (4):
  - Famcru Crs, Tygerberg Hills, Western Cape
  - Wits RHI Shandukani Research Centre CRS, Johannesburg
  - Soweto CRS, Site 8052, Soweto
  - Umlazi CRS, Umlazi
- Thailand (3):
  - Siriraj Hospital Mahidol University, Bangkok
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Uganda (2):
  - Baylor-Uganda CRS, Kampala
  - MU-JHU Care Limited CRS, Kampala

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- [Result] Gaur AH, Capparelli EV, Calabrese K, Baltrusaitis K, Marzinke MA, McCoig C, Van Solingen-Ristea RM, Mathiba SR, Adeyeye A, Moye JH, Heckman B, Lowenthal ED, Ward S, Milligan R, Samson P, Best BM, Harrington CM, Ford SL, Huang J, Crauwels H, Vandermeulen K, Agwu AL, Smith-Anderson C, Camacho-Gonzalez A, Ounchanum P, Kneebone JL, Townley E, Bolton Moore C; IMPAACT 2017 Collaborators; IMPAACT 2017 Team. Safety and pharmacokinetics of oral and long-acting injectable cabotegravir or long-acting injectable rilpivirine in virologically suppressed adolescents with HIV (IMPAACT 2017/MOCHA): a phase 1/2, multicentre, open-label, non-comparative, dose-finding study. Lancet HIV. 2024 Apr;11(4):e211-e221. doi: 10.1016/S2352-3018(23)00300-4. PMID 38538160
- [Result] Lowenthal ED, Chapman J, Ohrenschall R, Calabrese K, Baltrusaitis K, Heckman B, Yin DE, Agwu AL, Harrington C, Van Solingen-Ristea RM, McCoig CC, Adeyeye A, Kneebone J, Chounta V, Smith-Anderson C, Camacho-Gonzalez A, D'Angelo J, Bearden A, Crauwels H, Huang J, Buisson S, Milligan R, Ward S, Bolton-Moore C, Gaur AH; IMPAACT 2017 Collaborators; IMPAACT 2017 Team. Acceptability and tolerability of long-acting injectable cabotegravir or rilpivirine in the first cohort of virologically suppressed adolescents living with HIV (IMPAACT 2017/MOCHA): a secondary analysis of a phase 1/2, multicentre, open-label, non-comparative dose-finding study. Lancet HIV. 2024 Apr;11(4):e222-e232. doi: 10.1016/S2352-3018(23)00301-6. PMID 38538161
- [Derived] Gaur AH, Baltrusaitis K, Capparelli EV, Moye JH, Yin DE, Masheto G, Buisson S, Harrington CM, Marzinke MA, Lowenthal ED, Scheckter R, Ace A, Ward S, Milligan R, Whitson K, Huang J, Cheung SYA, Best BM, Townley E, Roberts G, Kakuda TN, Birmingham E, Mathiba SR, Aurpibul L, Korutaro V, Smith C, Patel F, Moodley E, Bolton-Moore C; IMPAACT 2017 Collaborators; IMPAACT 2017 Team. Safety, antiviral activity, and pharmacokinetics of long-acting injectable cabotegravir-rilpivirine in virologically suppressed adolescents living with HIV-1 (IMPAACT 2017/MOCHA): 48-week results of a multinational, phase 1/2, single-arm study. Lancet HIV. 2026 Jan 14:S2352-3018(25)00242-5. doi: 10.1016/S2352-3018(25)00242-5. Online ahead of print. PMID 41547359
- [Derived] Lowenthal ED, Chapman J, Baltrusaitis K, Kovic G, Merchant S, Branch K, Tsosie C, Vaca MZ, Heckman B, Van Solingen-Ristea RM, Harrington CM, Yin DE, Townley E, Whitton M, Agwu AL, Smith C, Paul ME, Violari A, Moodley E, Owor M, Chokephaibulkit K, Fry S, Jao J, Mitchell CD, Buisson S, Ace A, Kolobova I, Bolton-Moore C, Gaur AH; IMPAACT 2017 Collaborators; IMPAACT 2017 Team. Acceptability and tolerability of long-acting injectable cabotegravir-rilpivirine in adolescents with HIV-1 (IMPAACT 2017/MOCHA): 48-week results of a multicentre, open-label, non-comparative phase 1/2 trial. Lancet HIV. 2026 Jan 14:S2352-3018(25)00241-3. doi: 10.1016/S2352-3018(25)00241-3. Online ahead of print. PMID 41547358
- [Derived] Okesanya OJ, Ayeni RA, Amadin P, Ngwoke I, Amisu BO, Ukoaka BM, Ahmed MM, Oso TA, Musa SS, Lucero-Prisno DE. Advances in HIV Treatment and Vaccine Development: Emerging Therapies and Breakthrough Strategies for Long-Term Control. AIDS Res Treat. 2025 Jul 4;2025:6829446. doi: 10.1155/arat/6829446. eCollection 2025. PMID 40655875
- [Derived] Moore CB, Baltrusaitis K, Best BM, Moye JH, Townley E, Violari A, Heckman B, Buisson S, Van Solingen-Ristea RM, Capparelli EV, Marzinke MA, Lowenthal ED, Ward S, Krotje C, Milligan R, Agwu AL, Huang J, Cheung SYA, McCoig C, Yin DE, Roberts G, Crauwels H, Van Eygen V, Zabih S, Masheto G, Ounchanum P, Aurpibul L, Korutaro V, Gaur AH; IMPAACT 2017 Collaborators for the IMPAACT 2017 Team. Safety of combined long-acting injectable cabotegravir and long-acting injectable rilpivirine in virologically suppressed adolescents with HIV (IMPAACT 2017/MOCHA): a phase 1/2, multicentre, open-label, non-comparative, dose-finding study. Lancet HIV. 2025 Mar;12(3):e191-e200. doi: 10.1016/S2352-3018(24)00344-8. PMID 40049924
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: ICH Criteria for Meeting Serious Adverse Events — https://database.ich.org/sites/default/files/E2A_Guideline.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual for Cohort 1 occurred between April 2019 and November 2021 at 15 different medical clinic sites across Botswana, South Africa, Thailand, and the United States. Accrual for Cohort 2 occurred between July 2021 and August 2022 at 18 different medical clinic sites across Botswana, South Africa, Thailand, Uganda, and the United States.
Pre-assignment Details: 55 participants were enrolled into Cohort 1C/1R, and 44 of these participants continued to Cohort 2. An additional 100 participants enrolled into Cohort 2. Parents/caregivers (n = 13) are not included in the participant flow result section because no baseline measurements were collected for these participants. In addition, no data collected from these participants contributed to the reporting of results for primary or secondary objectives.
Groups:
- Cohort 1C: CAB: Step 1: CAB administered orally as one 30 mg tablet once daily, beginning at the Entry visit, for 4-6 weeks.
  Step 2 (Q4W dosing): CAB LA administered as three single intramuscular (IM) injections four weeks apart (600 mg injection at Week 4b, 400 mg injection at Week 8, and 400 mg injection at Week 12).
  Step 2 (Q8W dosing): CAB LA administered as two single IM injections four weeks apart (600 mg injection at Week 4b and 600 mg injection at Week 8).
  Oral Cabotegravir (CAB): 30 mg tablets administered orally
  Long-Acting Injectable Cabotegravir (CAB LA): Administered by intramuscular (IM) injection
  Combination Antiretroviral Therapy (cART): Participants continued their pre-study cART regimen. The antiretroviral drugs in participants' cART regimens were not provided through the study.
- Cohort 1R: RPV: Step 1: RPV administered orally as one 25 mg tablet once daily, beginning at the Entry visit, for 4-6 weeks.
  Step 2 (Q4W dosing): RPV LA administered as three single IM injections four weeks apart (900 mg injection at Week 4b, 600 mg injection at Week 8, 600 mg injection at and Week 12).
  Step 2 (Q8W dosing): RPV LA administered as two single IM injections four weeks apart (900 mg injection at Week 4b and 900 mg injection at Week 8).
  Oral Rilpivirine (RPV): 25 mg tablets administered orally
  Long-Acting Injectable Rilpivirine (RPV LA): Administered by intramuscular (IM) injection
  Combination Antiretroviral Therapy (cART): Participants continued their pre-study cART regimen. The antiretroviral drugs in participants' cART regimens were not provided through the study.
- Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA: Step 3: CAB administered orally as one 30 mg tablet once daily and RPV administered orally as one 25 mg tablet once daily, beginning at the Entry visit for 4-6 weeks.
  Step 4: First and second injections: CAB LA administered as a 600 mg IM injection and RPV LA administered as a 900 mg IM injection at Week 4b and at Week 8. Subsequent injections: starting at Week 16, CAB LA administered as a 600 mg IM injection and RPV LA administered as a 900 mg IM injection every eight weeks through Week 96 or final safety extension visit.
  Oral Cabotegravir (CAB): 30 mg tablets administered orally
  Oral Rilpivirine (RPV): 25 mg tablets administered orally
  Long-Acting Injectable Cabotegravir (CAB LA): Administered by intramuscular (IM) injection
  Long-Acting Injectable Rilpivirine (RPV LA): Administered by intramuscular (IM) injection
Period: Cohort 1 Treatment Initiation to Week 16
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 30 | 25 | 0 | 0
Completed | 29 | 23 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: Cohort 1 Week 16 Through End of Cohort 1
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 29 | 23 | 0 | 0
Completed | 28 | 21 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Cohort 2 Treatment Initiation to Week 24
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 0 (Cohort 1C participants who enrolled to Cohort 2 are counted within the Cohort 2A column.) | 0 (Cohort 1R participants who enrolled to Cohort 2 are counted within the Cohort 2A column.) | 144 | 0
Completed | 0 | 0 | 141 | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 1 | 0
Period: Cohort 2 Week 24 to Week 48
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 0 | 0 | 141 | 0
Completed | 0 | 0 | 140 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: Cohort 2 Week 48 to Week 96
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 0 | 0 | 140 | 0
Completed | 0 | 0 | 137 | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Cohort 2 Safety Extension
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA
Started | 0 | 0 | 117 (18 participants completed the study at Week 96, and 2 participants discontinued study treatment following the Week 96 visit.) | 0
Completed | 0 | 0 | 116 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who have taken at least 1 dose of any study product on the respective cohort. For participants enrolled in both Cohort 1 and Cohort 2, the baseline value summarized is from the corresponding cohort. Baseline characteristics for parents/caregivers are not reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA | Cohort 2B: CAB LA + RPV LA | Total
Number analyzed (Participants) | 30 | 25 | 144 | 0 | 199
Age, Continuous [Median (Full Range); unit: years] — Age is summarized as age at first enrollment to either Cohort 1 or Cohort 2. Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  years
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 | 15 [12 to 17] | 16 [12 to 17] |  |  | 15 [12 to 17]
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 |  |  | 15 [12 to 17] |  | 15 [12 to 17]
Age, Customized [Count of Participants; unit: Participants] — Age is summarized as age at first enrollment to either Cohort 1 or Cohort 2. Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: 12 | 1 | 3 |  | 0 | 4
    Cohort 1: 13 | 5 | 0 |  | 0 | 5
    Cohort 1: 14 | 7 | 3 |  | 0 | 10
    Cohort 1: 15 | 6 | 4 |  | 0 | 10
    Cohort 1: 16 | 4 | 4 |  | 0 | 8
    Cohort 1: 17 | 7 | 11 |  | 0 | 18
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: 12 |  |  | 11 |  | 11
    Cohort 2: 13 |  |  | 23 |  | 23
    Cohort 2: 14 |  |  | 19 |  | 19
    Cohort 2: 15 |  |  | 35 |  | 35
    Cohort 2: 16 |  |  | 27 |  | 27
    Cohort 2: 17 |  |  | 29 |  | 29
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: Female | 14 | 12 |  |  | 26
    Cohort 1: Male | 16 | 13 |  |  | 29
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: Female |  |  | 74 |  | 74
    Cohort 2: Male |  |  | 70 |  | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: Hispanic or Latino | 0 | 3 |  |  | 3
    Cohort 1: Not Hispanic or Latino | 30 | 22 |  |  | 52
    Cohort 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: Hispanic or Latino |  |  | 3 |  | 3
    Cohort 2: Not Hispanic or Latino |  |  | 141 |  | 141
    Cohort 2: Unknown or Not Reported |  |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Cohort 1: Asian | 9 | 0 |  |  | 9
    Cohort 1: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Cohort 1: Black or African American | 21 | 21 |  |  | 42
    Cohort 1: White | 0 | 4 |  |  | 4
    Cohort 1: More than one race | 0 | 0 |  |  | 0
    Cohort 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: American Indian or Alaska Native |  |  | 0 |  | 0
    Cohort 2: Asian |  |  | 36 |  | 36
    Cohort 2: Native Hawaiian or Other Pacific Islander |  |  | 0 |  | 0
    Cohort 2: Black or African American |  |  | 106 |  | 106
    Cohort 2: White |  |  | 2 |  | 2
    Cohort 2: More than one race |  |  | 0 |  | 0
    Cohort 2: Unknown or Not Reported |  |  | 0 |  | 0
Region of Enrollment, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: United States | 8 | 17 |  |  | 25
    Cohort 1: Botswana | 0 | 5 |  |  | 5
    Cohort 1: South Africa | 14 | 3 |  |  | 17
    Cohort 1: Uganda | 0 | 0 |  |  | 0
    Cohort 1: Thailand | 8 | 0 |  |  | 8
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: United States |  |  | 20 |  | 20
    Cohort 2: Botswana |  |  | 25 |  | 25
    Cohort 2: South Africa |  |  | 43 |  | 43
    Cohort 2: Uganda |  |  | 20 |  | 20
    Cohort 2: Thailand |  |  | 36 |  | 36
HIV-1 RNA [Count of Participants; unit: Participants] — The last available HIV-1 RNA viral load on or before the first dose of treatment for the corresponding cohort. Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants.
  Participants
    Cohort 1: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1: <50 copies/mL | 30 | 24 |  |  | 54
    Cohort 1: >=50 copies/mL | 0 | 1 |  |  | 1
    Cohort 2: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2: <50 copies/mL |  |  | 138 |  | 138
    Cohort 2: >=50 copies/mL |  |  | 6 |  | 6
Quality of Life Dimension Scores [Median (Inter-Quartile Range); unit: units on a scale] — Calculated dimension scores from the PedsQL: Pediatric Quality of Life Inventory range from 0 (worst) to 100 (best). Population: Baseline characteristics are reported separately for Cohort 1 and Cohort 2 participants. Questions used for School Functioning Dimension are only answered by participants who are attempting school at the time of the evaluation. One participant in Cohort 1R and 11 participants in Cohort 2 did not respond to these questions.
  units on a scale
    Cohort 1 Physical Functioning Dimension: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 Physical Functioning Dimension | 96.9 [93.8 to 100] | 100 [96.9 to 100] |  |  | 100 [93.8 to 100]
    Cohort 1 Emotional Functioning Dimension: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 Emotional Functioning Dimension | 90 [80 to 100] | 90 [70 to 100] |  |  | 90 [75 to 100]
    Cohort 1 Social Functioning Dimension: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 Social Functioning Dimension | 100 [90 to 100] | 95 [90 to 100] |  |  | 100 [90 to 100]
    Cohort 1 School Functioning Dimension: number analyzed (Participants) | 30 | 24 | 0 | 0 | 54
    Cohort 1 School Functioning Dimension | 80 [70 to 90] | 70 [60 to 87.5] |  |  | 80 [65 to 90]
    Cohort 1 Psychosocial Functioning Dimension: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 Psychosocial Functioning Dimension | 90 [81.7 to 96.7] | 83.3 [76.7 to 95] |  |  | 90 [78.3 to 95]
    Cohort 1 Total Functioning Dimension: number analyzed (Participants) | 30 | 25 | 0 | 0 | 55
    Cohort 1 Total Functioning Dimension | 92.9 [87 to 96.7] | 89.1 [83.7 to 95.7] |  |  | 91.3 [83.7 to 95.8]
    Cohort 2 Physical Functioning: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 Physical Functioning |  |  | 100 [93.8 to 100] |  | 100 [93.8 to 100]
    Cohort 2 Emotional Functioning Dimension: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 Emotional Functioning Dimension |  |  | 100 [85 to 100] |  | 100 [85 to 100]
    Cohort 2 Social Functioning Dimension: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 Social Functioning Dimension |  |  | 100 [90 to 100] |  | 100 [90 to 100]
    Cohort 2 School Functioning Dimension: number analyzed (Participants) | 0 | 0 | 133 | 0 | 133
    Cohort 2 School Functioning Dimension |  |  | 80 [70 to 90] |  | 80 [70 to 90]
    Cohort 2 Psychosocial Functioning: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 Psychosocial Functioning |  |  | 91.7 [83.3 to 96.7] |  | 91.7 [83.3 to 96.7]
    Cohort 2 Total Functioning: number analyzed (Participants) | 0 | 0 | 144 | 0 | 144
    Cohort 2 Total Functioning |  |  | 94.6 [84.8 to 97.8] |  | 94.6 [84.8 to 97.8]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Event (Cohort 1)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE through 4 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 4
Population: Cohort 1 Evaluable: Cohort 1 participants who were treated exclusively on the dose being evaluated for a given cohort, and either (1) completed all treatment regimen through Cohort 1 Week 4 and completed the Week 4 visit or (2) experienced any of the following: death attributable to the study product; study product-related Grade 3 or higher event (excluding injection site adverse events); OR permanently discontinued from treatment due to study product-related toxicity (regardless of grade).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 30
proportion of participants | 0 [0 to 0.12]

2. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE assessed as related by the site investigator of record to study product through 4 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 30
proportion of participants | 0 [0 to 0.12]

3. Primary Outcome: Proportion of Participants Who Had Serious Adverse Events Meeting International Conference on Harmonisation (ICH) Criteria Assessed as Related to Study Product/s (Cohort 1)
Description: Adverse events (AE) were assessed as a Serious AE by ICH criteria. Per ICH, a serious AE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect (see references for additional details). We present the proportion of participants with at least one serious AE assessed as related to study product by the site investigator of record through 4 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 30
proportion of participants | 0 [0 to 0.12]

4. Primary Outcome: Proportion of Participants Who Permanently Discontinued Study Product Due to Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: We present the proportion of participants who permanently discontinued study product due to adverse events (AEs) assessed as related to study product by the site investigator of record through 4 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 30
proportion of participants | 0 [0 to 0.12]

5. Primary Outcome: Proportion of Participants Who Died Due to Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: We present the proportion of participants who died due to adverse events assessed as related to study product by the site investigator of record through 4 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 30
proportion of participants | 0 [0 to 0.12]

6. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events (Cohort 1)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE through 16 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 16
Population: Cohort 1 Evaluable: Cohort 1 participants who were treated exclusively on the dose being evaluated for a given cohort, and either (1) completed all treatment regimen through Cohort 1 Week 16 and completed the Week 16 visit or (2) experienced any of the following: death attributable to the study product; study product-related Grade 3 or higher event (excluding injection site adverse events); OR permanently discontinued from treatment due to study product-related toxicity (regardless of grade)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0.24 [0.10 to 0.44] | 0.22 [0.07 to 0.44]

7. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE assessed as related to study product by the site investigator of record through 16 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 16
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0.035 [0.001 to 0.18] | 0.04 [0.001 to 0.22]

8. Primary Outcome: Proportion of Participants Who Had Serious Adverse Events Meeting International Conference on Harmonisation (ICH) Criteria Assessed as Related to Study Product/s (Cohort 1)
Description: Adverse events (AE) were assessed as a Serious AE by ICH criteria. Per ICH, a serious AE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect (see references for additional details). We present the proportion of participants with at least one serious AE assessed as related to study product by the site investigator of record through 16 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 16
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0 [0 to 0.12] | 0 [0 to 0.15]

9. Primary Outcome: Proportion of Participants Who Permanently Discontinued Study Product Due to Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: We present the proportion of participants who permanently discontinued study product due to adverse events (AEs) assessed as related to study product by the site investigator of record through 16 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 16
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0 [0 to 0.12] | 0.044 [0.001 to 0.22]

10. Primary Outcome: Proportion of Participants Who Died Due to Adverse Events Assessed as Related to Study Product/s (Cohort 1)
Description: We present the proportion of participants who died due to adverse events assessed as related to study product by the site investigator of record through 16 weeks post-treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 1 Treatment Initiation through Week 16
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0 [0 to 0.12] | 0 [0 to 0.15]

11. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events (Cohort 2)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE through 24 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 Treatment Initiation through Week 24
Population: Cohort 2 Naive Evaluable: Cohort 2 participants who did not participate in Cohort 1, were treated exclusively on the final recommended dose for Cohort 2, and either (1) completed all treatment regimens through Week 24 visit or (2) experienced any of the following: death attributable to the study product(s); study product(s)-related Grade 3 or higher event (excluding ISR AEs); OR permanently discontinued from treatment due to study product(s)-related toxicity during the dose-finding period.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0.10 [0.05 to 0.18]

12. Primary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE assessed as related to study product by the site investigator of record through 24 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 Treatment Initiation through Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0 [0 to 0.04]

13. Primary Outcome: Proportion of Participants Who Had Serious Adverse Events Meeting ICH Criteria Assessed as Related to Study Product/s (Cohort 2)
Description: Adverse events (AE) were assessed as a Serious AE by ICH criteria. Per ICH, a serious AE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect (see references for additional details). We present the proportion of participants with at least one serious AE assessed as related to study product by the site investigator of record through 24 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 Treatment Initiation through Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0 [0 to 0.04]

14. Primary Outcome: Proportion of Participants Who Permanently Discontinued Study Product Due to Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: We present the proportion of participants who permanently discontinued study product due to adverse events (AEs) assessed as related to study product by the site investigator of record through 24 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 Treatment Initiation through Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0 [0 to 0.04]

15. Primary Outcome: Proportion of Participants Who Died Due to Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: We present the proportion of participants who died due to adverse events assessed as related to study product by the site investigator of record through 24 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 Treatment Initiation through Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0 [0 to 0.04]

16. Primary Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve (AUC) for Step 1 Oral CAB (Cohort 1C)
Description: AUC calculated using non-compartmental methods with linear up-log down trapezoidal rule (Phoenix WinNonlin v 8.3, Certara®). We present the geometric mean of the AUC with associated geometric coefficient of variation.
Time Frame: Week 2: Samples collected pre-dose and 1, 2, 3, 4, 8, and (for Q4W dosing) 24 hours post-dose
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1 and had an available AUC measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ug)/mL
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 29
(h*ug)/mL | 139 (59.1)

17. Primary Outcome: Apparent Total Body Clearance (CL/F) of Step 1 Oral CAB (Cohort 1C)
Description: We present the geometric mean of the total body clearance of CAB and associated geometric coefficient of variation, based on analysis of intensive pharmacokinetic (PK) samples.
Time Frame: Week 2: Samples collected pre-dose and 1, 2, 3, 4, 8 and (for Q4W dosing) 24 hours post-dose
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1 and have an available total body clearance measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 29
mL/h | 216.0 (59.1)

18. Primary Outcome: Geometric Mean Maximum Plasma Concentration (Cmax) of Oral CAB (Cohort 1C)
Description: We present the geometric mean of the maximum plasma concentration of CAB and associated geometric coefficient of variation, based on analysis of intensive PK samples
Time Frame: Week 2: Samples collected pre-dose and 1, 2, 3, 4, 8 and (for Q4W dosing) 24 hours post-dose
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1 with an available Cmax measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 29
ug/mL | 8.90 (43.1)

19. Primary Outcome: Time of Maximum Concentration (Tmax) of Oral CAB (Cohort 1C)
Description: We present the mean time of maximum concentration of CAB and associated standard deviation, based on analysis of intensive PK samples.
Time Frame: Week 2: Samples collected pre-dose and 1, 2, 3, 4, 8, and (for Q4W dosing) 24 hours post-dose
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1 with an available Tmax measurement
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 29
h | 2.73 (1.13)

20. Primary Outcome: Geometric Mean Pre-dose Concentration (C0) of Oral CAB (Cohort 1C)
Description: We present the geometric mean pre-dose CAB concentration and associated geometric coefficient of variation, based on analysis of intensive PK samples.
Time Frame: Week 2: Samples collected pre-dose and 1, 2, 3, 4, 8, and (for Q4W dosing) 24 hours post-dose
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1 with an available pre-dose concentration measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB
Number analyzed (Participants) | 29
ug/mL | 4.09 (96.1)

21. Primary Outcome: Geometric Mean Concentration of LA CAB/LA RPV at Week 16 (Cohort 1 Q4W)
Description: We present the geometric mean concentration of LA CAB/LA RPV and associated geometric coefficients of variation for participants on the Q4W dosing regimen, based on analysis of pre-dose PK sample.
Time Frame: Week 16
Population: Cohort 1 Q4W: Cohort 1 participants who received the Q4W dosing regimen on Cohort 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 8 | 12
ug/mL | 2.91 (58.8) | 0.0644 (59.9)

22. Primary Outcome: Geometric Mean Maximum Plasma Concentration (Cmax) of LA CAB/LA RPV (Cohort 1 Q4W)
Description: We present the geometric mean of the maximum plasma concentration of LA CAB/LA RPV and associated geometric coefficient of variation for the first injection in participants on the Q4W dosing regimen, based on analysis of intensive PK samples.
Time Frame: Samples collected at Weeks 4b, 5, 6, and 8
Population: Cohort 1 Q4W: Cohort 1 participants who received the Q4W dosing regimen on Cohort 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 8 | 13
ug/mL | 9.56 (32.2) | 0.132 (35.5)

23. Primary Outcome: Time of Maximum Concentration (Tmax) of LA CAB/LA RPV (Cohort 1 Q4W)
Description: We present the mean time of maximum concentration of LA CAB/LA RPV at the first injection and associated standard deviation for participants on the Q4W dosing regimen, based on analysis of intensive PK samples.
Time Frame: Samples collected at Weeks 4b, 5, 6, 8
Population: Cohort 1 participants who received the Q4W dosing regimen on Cohort 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 8 | 13
h | 1.50 (0.551) | 89.6 (162)

24. Primary Outcome: Geometric Mean Pre-dose Concentration (C0) of LA CAB/LA RPV (Cohort 1 Q4W)
Description: We present the geometric mean pre-dose concentrations of each injection and associated geometric coefficient of variation for participants on the Q4W dosing regimen, based on analysis of pre-dose PK samples.
Time Frame: Week 4b, Week 8, Week 12
Population: Cohort 1 participants who received the Q4W dosing regimen on Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Cohort 1R: RPV: Step 1: RPV administered orally as one 25 mg tablet once daily, beginning at the Entry visit, for 4-6 weeks.
  Step 2 (Q4W dosing): RPV LA administered as three single IM injections four weeks apart (900 mg injection at Week 4b, 600 mg injection at Week 8, 600 mg injection at and Week 12).
  Step 2 (Q8W dosing): RPV LA administered as two single IM injections four weeks apart 900 mg injection at Week 4b and (900 mg injection at Week 8).
  Oral Rilpivirine (RPV): 25 mg tablets administered orally
  Long-Acting Injectable Rilpivirine (RPV LA): Administered by intramuscular (IM) injection
  Combination Antiretroviral Therapy (cART): Participants continued their pre-study cART regimen. The antiretroviral drugs in participants' cART regimens were not provided through the study.
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 8 | 13
ug/mL
  Week 4b | 5.46 (39.6) | 0.0704 (227)
  Week 8 | 2.10 (37.0) | 0.0441 (75.9)
  Week 12 | 2.73 (76.7) | 0.0555 (56.7)

25. Primary Outcome: Geometric Mean Concentration of LA CAB/LA RPV at Week 16 (Cohort 1 Q8W)
Description: We present the geometric mean concentration of LA CAB/LA RPV and associated geometric coefficients of variation for participants on the Q4W dosing regimen, based on analysis of the pre-dose PK sample.
Time Frame: Week 16
Population: Cohort 1 participants who received the Q8W dosing regimen on Cohort 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 21 | 10
ug/mL | 1.01 (237) | 0.0449 (38.2)

26. Primary Outcome: Geometric Mean Maximum Plasma Concentration (Cmax) of LA CAB/LA RPV (Cohort 1 Q8W)
Description: We present the geometric mean of the maximum plasma concentration of LA CAB/LA RPV and associated geometric coefficient of variation for the first injection in participants on the Q8W dosing regimen, based on analysis of intensive PK samples.
Time Frame: Samples collected at Weeks 4b, 5, and 8
Population: Cohort 1 participants who received the Q8W dosing regimen on Cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 21 | 10
ug/mL | 6.42 (42.2) | 0.129 (39.4)

27. Primary Outcome: Time of Maximum Concentration (Tmax) of LA CAB/LA RPV (Cohort 1 Q8W)
Description: We present the mean time of maximum concentration of LA CAB/LA RPV at the first injection and associated standard deviation for participants on the Q8W dosing regimen, based on analysis of intensive PK samples.
Time Frame: Samples collected at Weeks 4b, 5, and 8
Population: Cohort 1 participants who received the Q8W dosing regimen on Cohort 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 21 | 10
h | 1.84 (0.829) | 18.6 (53.5)

28. Primary Outcome: Geometric Mean Pre-dose Concentration (C0) of LA CAB/LA RPV (Cohort 1 Q8W)
Description: We present the geometric mean pre-dose concentration of the first injection and associated geometric coefficient of variation for participants on the Q4W dosing regimen, based on analysis of pre-dose PK samples.
Time Frame: Week 4b, Week 8
Population: We present the geometric mean pre-dose concentration of the first injection and associated coefficient of variation for participants on the Q4W dosing regimen, based on analysis of intensive PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 21 | 10
ug/mL
  Week 4b | 2.89 (194) | 0.0703 (24.8)
  Week 8 | 1.33 (105) | 0.0327 (28.8)

29. Secondary Outcome: Proportion of Participants With HIV-1 RNA < 50 Copies/mL (Cohort 1)
Description: We present the proportion of participants with results of HIV-1 RNA < 50 copies/mL at Week 16
Time Frame: Week 16
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1
Measure: Number; unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 28 | 22
proportion of participants | 0.964 | 1.00

30. Secondary Outcome: Proportion of Participants Who Reported "Hurts Whole Lot" or "Hurts Worst" in Regards to Being Bothered by Pain During Injection of CAB LA or RPV LA (Cohort 1)
Description: Results collected via administration of Pain During Injection survey to participants after receiving injection. Pain during injections was assessed using the Faces Pain Scale-Revised which includes 6 visual and text options: "no hurt," "hurts little bit," "hurts little more," "hurts even more," "hurts whole lot" and "hurts worst".
Time Frame: Week 8
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1
Measure: Number; unit: proportion of participants
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
proportion of participants | 0 | 0.043

31. Secondary Outcome: Median Dimension of Quality of Life Scores
Description: A commonly used 23-item Pediatric Quality of Life Inventory, the PedsQLTM, was used to measure physical, emotional, and social dimensions of health as well as school functioning. Question responses were used to generate scores from 0-100 (100 being the best quality of life) based on the PedsQLTM guidelines. The number of participants drops slightly for the school functioning result as not all participants are eligible to answer these school-related questions.
Time Frame: Week 16
Population: Cohort 1 All Treated: Cohort 1 participants who have taken at least 1 dose of any study product on Cohort 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV
Number analyzed (Participants) | 29 | 23
score on a scale
  Physical Functioning | 96.9 [90.6 to 100] | 100 [93.8 to 100]
  Emotional Functioning | 95 [80 to 100] | 95 [90 to 100]
  Social Functioning | 100 [95 to 100] | 100 [95 to 100]
  School Functioning | 80 [65 to 90] | 85 [80 to 95]
  Psychosocial Functioning | 91.7 [76.7 to 96.7] | 91.7 [86.7 to 96.7]
  Total Functioning | 93.5 [82.6 to 96.7] | 94.6 [90.2 to 97.8]

32. Secondary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events (Cohort 2)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE through 48 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 treatment initiation through Week 48
Population: Cohort 2 Naive Evaluable: Cohort 2 participants who did not participate in Cohort 1, were treated exclusively on the final recommended dose for Cohort 2, and either (1) completed all treatment regimens through Week 48 visit or (2) experienced any of the following: death attributable to the study product(s); study product(s)-related Grade 3 or higher event (excluding ISR AEs); OR permanently discontinued from treatment due to study product(s)-related toxicity during the treatment period.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0.14 [0.08 to 0.23]

33. Secondary Outcome: Proportion of Participants Who Had Grade 3 or Higher Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an adverse event (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE assessed as related to study product by the site investigator of record through 48 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 treatment initiation through Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0.02 [0.003 to 0.07]

34. Secondary Outcome: Proportion of Participants Who Had Serious Adverse Events Meeting ICH Criteria, as Cited in References, Assessed as Related to Study Product/s (Cohort 2)
Description: Adverse events (AE) were assessed as a Serious AE by ICH criteria. Per ICH, a serious AE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect (see references for additional details). We present the proportion of participants with at least one serious AE assessed as related to study product by the site investigator of record through 48 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 treatment initiation through Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0 [0 to 0.04]

35. Secondary Outcome: Proportion of Participants Who Permanently Discontinued Study Product Due to Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: We present the proportion of participants who permanently discontinued study product due to adverse events (AEs) assessed as related to study product by the site investigator of record through 48 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 treatment initiation through Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0 [0 to 0.04]

36. Secondary Outcome: Proportion of Participants Who Died Due to Adverse Events Assessed as Related to Study Product/s (Cohort 2)
Description: We present the proportion of participants who died due to adverse events assessed as related to study product by the site investigator of record through 48 weeks post-Cohort 2 treatment initiation, bounded by an exact 95% confidence interval (CI).
Time Frame: Cohort 2 treatment initiation through Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0 [0 to 0.04]

37. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA >= 50 Copies/mL Per the FDA Snapshot (Cohort 2)
Description: We present the proportion of participants with HIV-1 RNA >= 50 copies/mL and associated exact 95% CI (Clopper-Pearson) per the FDA snapshot, based on laboratory evaluations.
Time Frame: Week 24
Population: Cohort 2 Naive Evaluable: Cohort 2 participants who did not participate in Cohort 1, were treated exclusively on the final recommended dose for Cohort 2, and either (1) completed all treatment regimens through Week 24 visit or (2) experienced any of the following: death attributable to the study product(s); study product(s)-related Grade 3 or higher event (excluding ISR AEs); OR permanently discontinued from treatment due to study product(s)-related toxicity during the treatment period
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0.02 [0.002 to 0.07]

38. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA >= 200 Copies/mL Per the FDA Snapshot (Cohort 2)
Description: We present the proportion of participants with HIV-1 RNA >= 200 copies/mL and associated exact 95% CI (Clopper-Pearson) per the FDA snapshot, based on laboratory evaluations.
Time Frame: Week 24
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 98
proportion of participants | 0 [0 to 0.037]

39. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA >= 50 Copies/mL Per the FDA Snapshot (Cohort 2)
Description: as for outcome 37
Time Frame: Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0 [0 to 0.04]

40. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA >= 200 Copies/mL Per the FDA Snapshot (Cohort 2)
Description: as for outcome 38
Time Frame: Week 48
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 97
proportion of participants | 0 [0 to 0.04]

41. Secondary Outcome: Geometric Mean Pre-dose Concentration (C0) of Oral CAB and Oral RPV (Cohort 2)
Description: We present the geometric mean of the pre-dose concentration of oral CAB and oral RPV and associated coefficient of variation, based on analysis of pre-dose PK sample.
Time Frame: Week 2
Population: Cohort 2 All Treated: Cohort 2 participants who have taken at least 1 dose of any study product on Cohort 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 144
ug/mL
  CAB concentration | 6.65 (42.3)
  RPV concentration | 0.0708 (59.0)

42. Secondary Outcome: Geometric Mean Ratio of Pre-dose CAB and RPV Concentrations at Week 24: Pre-dose CAB and RPV Concentrations at Week 8 (Cohort 2)
Description: We present the geometric mean of the ratios of pre-dose CAB and RPV concentrations at Week 24:Week 8 and associated coefficient of variation, based on analysis of pre-dose PK samples.
Time Frame: Week 8 and Week 24
Population: Cohort 2 All Treated: Cohort 2 participants who have taken at least 1 dose of any study product on Cohort 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 139
ratio
  CAB Ratio | 1.14 (107)
  RPV Ratio | 1.35 (47.1)

43. Secondary Outcome: Geometric Mean Ratio of Pre-dose CAB and RPV Concentrations at Week 24: Pre-dose CAB and RPV Concentrations at Week 16 (Cohort 2)
Description: We present the geometric mean of the ratios of pre-dose CAB and RPV concentrations at Week 24:Week 16 and associated coefficient of variation, based on analysis of pre-dose PK samples.
Time Frame: Week 16 and Week 24
Population: Cohort 2 All Treated: Cohort 2 participants who have taken at least 1 dose of any study product on Cohort 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 139
ratio
  CAB Ratio | 0.974 (47.0)
  RPV Ratio | 1.22 (32.7)

44. Secondary Outcome: Geometric Mean Ratio of Pre-dose CAB and RPV Concentrations at Week 48: Pre-dose CAB and RPV Concentrations at Week 8 (Cohort 2)
Description: We present the geometric mean of the ratios of pre-dose CAB and RPV concentrations at Week 48:Week 8 and associated coefficient of variation, based on analysis of pre-dose PK samples.
Time Frame: Week 8 and Week 48
Population: Cohort 2 All Treated: Cohort 2 participants who have taken at least 1 dose of any study product on Cohort 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 138
ratio
  CAB Ratio | 1.31 (97.6)
  RPV Ratio | 1.84 (47.1)

45. Secondary Outcome: Geometric Mean Ratio of Pre-dose CAB and RPV Concentrations at Week 48: Pre-dose CAB and RPV Concentrations at Week 16 (Cohort 2)
Description: We present the geometric mean of the ratios of pre-dose CAB and RPV concentrations at Week 48:Week 16 and associated coefficient of variation, based on analysis of pre-dose PK samples.
Time Frame: Week 16 and Week 48
Population: Cohort 2 All Treated: Cohort 2 participants who have taken at least 1 dose of any study product on Cohort 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
Number analyzed (Participants) | 138
ratio
  CAB Ratio | 1.12 (50.9)
  RPV Ratio | 1.68 (37.9)

ADVERSE EVENTS:
Time Frame: Cohort 1: study entry through final study visit (Week 16, premature discontinuation prior to Week 16, final long-term safety follow-up visit, or Cohort 2 entry) Cohort 2: study entry through final study visit (Week 96, premature discontinuation prior to Week 96, final long-term safety follow-up visit, or final safety extension visit)
Description: According to the study protocol, safety outcome measures are summarized for Cohort 1C and Cohort 1R without respect to the dosing regimen. These adverse events are also presented by Cohort, and not by dosing regimen. Dosing regimen is only reported for PK related outcome measures and results. Adverse events were not collected for enrolled parent/caregivers in either Cohort 1 or Cohort 2.
Arm/Group | Cohort 1C: CAB | Cohort 1R: RPV | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25 | 0/144
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/25 | 9/144
Other Adverse Events (participants affected / at risk) | 28/30 | 23/25 | 136/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1C: CAB (N=30) | Cohort 1R: RPV (N=25) | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA (N=144)
Cataract (Eye disorders) | 0 | 0 | 1
Gastritis alcoholic haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1C: CAB (N=30) | Cohort 1R: RPV (N=25) | Cohort 2A: Oral CAB + Oral RPV and CAB LA + RPV LA (N=144)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 5
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 7
Sickle cell trait (Congenital, familial and genetic disorders) | 0 | 1 | 1
Ear canal erythema (Ear and labyrinth disorders) | 1 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 2
Ear pruritus (Ear and labyrinth disorders) | 0 | 2 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 2 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1
Noninfective myringitis (Ear and labyrinth disorders) | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 2
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Conjunctival pallor (Eye disorders) | 1 | 0 | 4
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 4
Eyelid oedema (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 4
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 2
Visual impairment (Eye disorders) | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 9
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 6
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 2
Breath odour (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 9
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2
Enlarged uvula (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1
Malpositioned teeth (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 11
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 2
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 6
Vomiting (Gastrointestinal disorders) | 1 | 4 | 12
Asthenia (General disorders) | 0 | 1 | 6
Chest discomfort (General disorders) | 2 | 2 | 4
Chills (General disorders) | 1 | 0 | 6
Complication of device insertion (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 8
Immediate post-injection reaction (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 1
Injection site hypoaesthesia (General disorders) | 0 | 1 | 1
Injection site induration (General disorders) | 0 | 0 | 3
Injection site joint pain (General disorders) | 0 | 0 | 1
Injection site nodule (General disorders) | 0 | 1 | 6
Injection site pain (General disorders) | 9 | 9 | 57
Injection site pruritus (General disorders) | 0 | 0 | 2
Injection site swelling (General disorders) | 1 | 1 | 8
Malaise (General disorders) | 0 | 0 | 3
Medical device pain (General disorders) | 0 | 0 | 1
Mucosal discolouration (General disorders) | 0 | 0 | 1
Mucosal disorder (General disorders) | 0 | 1 | 1
Mucosal hyperaemia (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 10
Pain (General disorders) | 1 | 0 | 4
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 26
Suprapubic pain (General disorders) | 0 | 0 | 1
Swelling face (General disorders) | 0 | 1 | 1
Vaccination site pain (General disorders) | 1 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 1 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 2 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 11
Conjunctivitis (Infections and infestations) | 0 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 1
Dermatophytosis (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 4
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 1
Herpes simplex pharyngitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 3
Injection site abscess (Infections and infestations) | 0 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 1
Latent syphilis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Malaria (Infections and infestations) | 0 | 0 | 7
Mumps (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 14
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 6
Otitis media (Infections and infestations) | 0 | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 0 | 2
Paronychia (Infections and infestations) | 0 | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 3
Plasmodium falciparum infection (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1
Proctitis gonococcal (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1
Scabies (Infections and infestations) | 0 | 0 | 1
Secondary syphilis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 3
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Syphilis genital (Infections and infestations) | 0 | 1 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 2
Typhoid fever (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 30
Urethritis (Infections and infestations) | 0 | 0 | 1
Urethritis gonococcal (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 7
Viral infection (Infections and infestations) | 0 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 10
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 3
Adverse event following immunisation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Perineal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 4
Product administration error (Injury, poisoning and procedural complications) | 0 | 0 | 2
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 4
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 2
Traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 19
Blood creatinine increased (Investigations) | 1 | 0 | 2
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 1 | 0 | 3
Blood pressure increased (Investigations) | 6 | 0 | 23
Blood pressure systolic increased (Investigations) | 1 | 0 | 15
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 2 | 1 | 7
Electrocardiogram PR prolongation (Investigations) | 1 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 2 | 0 | 9
Lipase increased (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 5
Platelet count decreased (Investigations) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 5
Weight increased (Investigations) | 0 | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 2
Underweight (Metabolism and nutrition disorders) | 2 | 0 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 9
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Delayed sleep phase (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 10
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 8 | 42
Migraine (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Sleep paralysis (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2
Speech disorder (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 4
Major depression (Psychiatric disorders) | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 3
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Breast discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2 | 5
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 52
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung hypoinflation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 28
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal mucosal discolouration (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Nasal mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 29
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 14
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 26
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dilated pores (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Physical assault (Social circumstances) | 0 | 0 | 1
Sexual abuse (Social circumstances) | 0 | 1 | 1
Substance use (Social circumstances) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 0 | 6
Hypotension (Vascular disorders) | 0 | 0 | 2
Pallor (Vascular disorders) | 0 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (4):
  • Study Protocol: V4.0 (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03497676/Prot_000.pdf
  • Study Protocol: V3.0 (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03497676/Prot_001.pdf
  • Statistical Analysis Plan: V2.0 (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03497676/SAP_002.pdf
  • Statistical Analysis Plan: V3.1 (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03497676/SAP_003.pdf